CLINICAL TRIAL: NCT04859803
Title: Efficacy of Rhomboid Intercostal Block With Sub-serratus Block on Perioperative Analgesia in Patients Undergoing Gynecomastia Surgery
Brief Title: Rhomboid Intercostal and Sub-serratus Block
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N-30-2021
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Rhomboid Intercostal Block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RISS group (Active Comparator): patients will receive rhomboid intercostal block under ultrasound guidance.
  Interventions: Procedure: Patients will be received rhomboid intercostal block under ultrasound guidance.
- Control group (Active Comparator): Patients will received the conventional intravenous analgesia
  Interventions: Drug: conventional intravenous analgesia

INTERVENTIONS:
Procedure: Patients will be received rhomboid intercostal block under ultrasound guidance. — Following endotracheal intubation, patients allotted to the RIB group were positioned in the lateral decubitus position with the chest on the operating side lying superiorly. The ipsilateral arm was abducted from the chest to move the scapula laterally. The RIB was performed as described previously [8]. A high-frequency (6-12 MHz) linear ultrasound probe (LOGIQ e ultrasonic system, Deutschland GmbH & Co. KG, Solingen, Germany) was placed medial to the medial border of the scapula in the oblique sagittal plane. The landmarks, i.e., the trapezius muscle, rhomboid muscle, intercostal muscles, pleura, and lung, were identified in the ultrasound. Under aseptic conditions, an 80-mm 21-gauge needle was inserted at the level of T6-7 in the ultrasound view. A single dose of 30 ml 0.25% bupivacaine will be injected in the interfascial plane between the rhomboid major and intercostal muscles. The spread of the local anesthetic solution under the rhomboid muscle was visualized by ultrasonography.
  Arms: RISS group
Drug: conventional intravenous analgesia — Following endotracheal intubation, patients will be received morphine sulfate (0.02 mg/kg) bolus doses were used to preserve MAP and HR within 20% of pre-induction readings
  Arms: Control group

SUMMARY:
The rhomboid intercostal block (RIB) can provide good analgesia effects after thoracic surgery . The ultrasound-guided RIB is novel analgesic techniques recently described by Elsharkawy et al. . Additionally, the RISS block anesthetizes the lateral cutaneous branches of the thoracic intercostal nerves and can be used in multiple clinical settings for chest wall and upper abdominal analgesia. However, the analgesic effects of the RISS block after breast surgery have not been analyzed through a randomized-controlled trial.

ELIGIBILITY:
Inclusion criteria Adult patients between 18-50 years. ASA physical status I and II Male gender

Exclusion criteria Patient refusal Contraindications to regional anesthesia Known allergy to local anesthetics Bleeding disorders Use of any anti-coagulants Inability to provide informed consent ASA III-IV

-

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 24 hours
  Postoperative morphine consumption

SECONDARY OUTCOMES:
recovery time | 1 hour
  The time from stopping anaesthetic agent until extubation
Pain evaluation | 24 hous
  Pain evaluation using the visual analog scale score,, 0= pain , 10= sever pain
time to first analgesia | 24 hous
  duration of block

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still work